CLINICAL TRIAL: NCT01835977
Title: Multi-Center Randomized Clinical Two Arm Intervention Study Evaluating Irreversible Electroporation for the Ablation of Localized Prostate Cancer
Brief Title: Multi-Center Randomized Clinical Trial Irreversible Electroporation for the Ablation of Localized Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinical Research Office of the Endourological Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013249
Record Dates: First submitted 2013-04-08; First posted 2013-04-19 (Estimated); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
Keywords: Focal therapy; Irreversible electroporation; Unilateral prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Focal ablation (Active Comparator): Focal ablation of unilateral histopathologically confirmed, organ confined prostate cancer using IRE
  Interventions: Device: Irreversible Electroporation (Nanoknife)
- Extended ablation (Active Comparator): Extended ablation unilateral histopathologically confirmed, organ confined prostate cancer using IRE
  Interventions: Device: Irreversible Electroporation (Nanoknife)

INTERVENTIONS:
Device: Irreversible Electroporation (Nanoknife)
  Other Names: Nanoknife

SUMMARY:
Multi-centre Randomized Clinical Trial: 106 patients with confirmed unilateral high-volume low risk (Gleason score 3 + 3) or intermediate risk prostate cancer (Gleason score 3 + 4) will undergo an IRE treatment. These patients will be randomized into one of the two groups of the study.

Group 1: Focal ablation of the prostate at the side of the positive biopsies (focal-ablation) Group 2: Extended ablation of the prostate (extended ablation)

Patients will have an ultrasound of the prostate and the imaging data will be entered into the Planning Software system of the IRE-device. The volume of the prostate is measured and a specified ablation zone will be determined. The patients will be admitted for overnight stay in the hospital on the morning of the scheduled IRE procedure. The IRE will be performed under general anaesthetic and the specified zone identified in the planning stage will be ablated. Two to four IRE electrode needles will be placed into the prostate under ultrasound image guidance with a perineal approach using a brachytherapy grid. When the needles are in place, electric pulses of one to two minutes duration are used to ablate the specified zone. The total procedure time will be approximately 1 hour.

Safety data will be collected and patients will be followed up at 1 day post-operatively, 1 month, 3 months, 6 months and 1, 2 and 3 year(s) post IRE.

ELIGIBILITY:
Inclusion Criteria

1. Histologically confirmed organ-confined unilateral prostate cancer with adjacent positive biopsies on transperineal template prostate biopsies or MRI targeted biopsies in combination with systematic biopsies (clinical stage T1c-T2b)
2. Gleason sum score 6 or 7
3. PSA <15 ng/ml or PSA > 15 ng/mL counselled with caution
4. Life expectancy of > 10 years

Exclusion Criteria

1. Bleeding disorder as determined by prothrombin time (PT) > 14.5 seconds, partial thromboplastin time (PTT) > 34 seconds, and Platelet Count < 140/uL
2. No ability to stop anticoagulant or anti-platelet therapy for 7 days prior the procedure.
3. Active urinary tract infection (UTI)
4. History of bladder neck contracture
5. Anaesthesia Surgical Assignment category IV or greater
6. History of inflammatory bowel disease
7. Concurrent major debilitating illness
8. Prior or concurrent malignancy except for basal cell carcinoma of the skin
9. Cardiac history including arrhythmias, ICD or pacemaker
10. Prostate calcifications greater than 5 mm.
11. Biologic or chemotherapy for prostate cancer
12. Hormonal therapy for prostate cancer within 6 months prior to procedure
13. Previous radiation to pelvis
14. Transurethral resection of the prostate / Urethral stent
15. Prior major rectal surgery (except haemorrhoids)

Ages: 50 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-06; Primary Completion 2020-01-30 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Patient experience (side-effects and quality of life) after IRE ablation of prostate cancer | 5 years
  To determine post procedural side-effects and Quality of life measured by International Prostate Symptom Score (IPSS), International Index of Erectile Function (IIEF) and Functional Assessment of Cancer Therapy-Prostate (FACT-P).

SECONDARY OUTCOMES:
Oncological efficacy IRE ablation of prostate cancer. | 5 years
  To determine if IRE focal ablation procedure is as effective as extended ablation measured by PSA, standardised transrectal biopsies and MRI findings in follow-up.
  To determine accurateness of ablation zone detection by MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Jean de la Rosette, MD, PhD, Study Chair — Clinical Research Office of the Endourological Society

REFERENCES:
- [Derived] Zhang K, Teoh J, Laguna P, Dominguez-Escrig J, Barret E, Ramon-Borja JC, Muir G, Bohr J, de Reijke TM, Pelechano Gomez P, Ng CF, Sanchez-Salas R, de la Rosette J. Effect of Focal vs Extended Irreversible Electroporation for the Ablation of Localized Low- or Intermediate-Risk Prostate Cancer on Early Oncological Control: A Randomized Clinical Trial. JAMA Surg. 2023 Apr 1;158(4):343-349. doi: 10.1001/jamasurg.2022.7516. PMID 36723911
- [Derived] Scheltema MJ, van den Bos W, de Bruin DM, Wijkstra H, Laguna MP, de Reijke TM, de la Rosette JJ. Focal vs extended ablation in localized prostate cancer with irreversible electroporation; a multi-center randomized controlled trial. BMC Cancer. 2016 May 5;16:299. doi: 10.1186/s12885-016-2332-z. PMID 27150293
- See also: Related Info — http://www.croesoffice.org